CLINICAL TRIAL: NCT00287677
Title: Double Strategy to Induce and Expand the T Cell Repertoire by the Administration of Growth Hormone and Vaccination in HIV-1 Infected Patients
Brief Title: Induction and Expansion of T Cell Repertoire Using Growth Hormone and Vaccination in HIV-1 Infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Hospital General Universitario Gregorio Marañon (Other); Carlos III Health Institute (Other Government)
Responsible Party: Germans Trias i Pujol Hospital, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIHCREC01
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2009-11-04 (Estimated); Status verified 2009-11

CONDITIONS: HIV Infections
Keywords: Growth Hormone; HIV-1; Vaccination; Thymopoiesis; HIV-specific responses; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Growth Hormone; Vaccination; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): growth hormone + vaccination + HAART
  Interventions: Biological: recombinant human Growth Hormone; Biological: Vaccination; Drug: HAART
- B (Experimental): growth hormone + HAART
  Interventions: Biological: recombinant human Growth Hormone; Drug: HAART
- C (Experimental): vaccination + HAART
  Interventions: Biological: Vaccination; Drug: HAART
- D (Active Comparator): control healthy HIV negative + vaccination
  Interventions: Biological: Vaccination

INTERVENTIONS:
Biological: recombinant human Growth Hormone — Growth Hormone during 6 months (30UG/KG/DAY)
  Arms: A; B
Biological: Vaccination — Vaccination (Hepatitis A+B + tetanus toxoid) at week 16
  Arms: A; C; D
Drug: HAART — HAART all over the trial
  Arms: A; B; C

SUMMARY:
Concomitant administration of recombinant human growth hormone (rhGH) may boost the expansion of immune reconstitution and broaden specific T cell responses not achievable by vaccination alone. The main objective of that study is to test the validity of this hypothesis with vaccines which are routinely administered to HIV-1 patients(tetanus toxoid and hepatitis A virus vaccines) in order to, if proven of value, use this strategy of HIV vaccination in the near future. This is a pilot, randomized, clinical open label study aimed to investigate thymic functionality and the HIV-specific responses after administration of rhGH in HIV-1 infected patients in highly active antiretroviral therapy (HAART) regimen.

DETAILED DESCRIPTION:
The purpose of a therapeutic vaccine is to control, induce and expand humoral and cellular immune responses capable to control HIV infection. The administration of a conventional vaccine results in the expansion of peripheral clones. Concomitant administration of rhGH may boost this expansion and reconstitute specific T cell responses not achievable by vaccination alone. In this study we want to investigate whether the administration of rhGH expand T cell repertoire and whether there is an increase in the specific cellular responses to HIV-1 and recall antigens and, lately, whether this responses can be further amplified after immunization with tetanus toxoid and hepatitis A vaccines. This Hypothesis will be evaluated by the measurement of thymic volume, the expansion of naïve, memory and effector cell subsets, analysis of thymic emigrants (TRECs) before, during and after rhGH administration and vaccination. Moreover, T cell receptor rearrangement, specific antibodies and cellular responses to antigenic peptides will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 asymptomatic patients in HAART regimen (> 6 months)
2. Viral load < 50 copies/ml
3. Number CD4 cells > 250 cells/mm3
4. Non responders to vaccination (tetanus toxoid and/or Hepatitis A virus)
5. Well-disposition to rhGh daily administration (6 months of treatment)

Exclusion Criteria:

1. AIDS outbreak
2. Allergy or hyperreactivity to rhGH or vaccines
3. Diabetes Mellitus
4. Renal, hepatic, pancreatic disorders
5. Chronic diseases
6. Dementia
7. Pregnancy

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2006-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients HIV+ that recover the immunospecific responses against tetanus toxoid and Hepatitis A at 24 weeks of rhGH administration (time of treatment interruption). | from 24 weeks post rhGH administration

SECONDARY OUTCOMES:
The rhGH activates the thymic function. | from one year post rhGH administration
This effect is lasting once the rhGH administration is interrupted. | from at least one year since the last rhGH administration

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventura Clotet, PhD, Study Director — IrsiCaixa Foundation-Germans Trias i Pujol Hospital; Lidia Ruiz, PhD, Principal Investigator — Irsicaixa Foundation-Germans Trias i Pujol Hospital; Jose Mª Gatell, PhD, Study Director — Hospital Clinic of Barcelona; Margarita Bofill, PhD, Study Director — Irsicaixa Foundation- Germans Trias i Pujol Hospital
Locations (2):
- Spain (2):
  - Germans Trias i Pujol Hospital, Badalona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona